CLINICAL TRIAL: NCT04320602
Title: Phase 4, Single-Arm Study of Ravulizumab in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria Currently Treated With High-Dose Eculizumab
Brief Title: Ravulizumab in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria Currently Treated With High-Dose Eculizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-401; 2019-003440-74 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-07

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PNH; Ravulizumab; Ultomiris; Eculizumab; Soliris
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab; ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): Participants will receive eculizumab during the 3-month Screening Period. Participants will then switch over to and receive weight-based doses of ravulizumab for the duration of the study Treatment Period (351 days).
  Interventions: Biological: Eculizumab; Biological: Ravulizumab

INTERVENTIONS:
Biological: Eculizumab — Participants must have been prescribed and be receiving a stable dose of eculizumab 1200 milligrams (mg) every 2 weeks (q2w) for at least 3 months prior to the Screening Period. During the Screening Period, participants will continue to receive eculizumab 1200 mg q2w.
  Other Names: Soliris
Biological: Ravulizumab — During the Treatment Period, participants will receive a loading dose of ravulizumab on Day 1, followed by maintenance doses on Day 15 and every 8 weeks, administered by intravenous infusion. Ravulizumab loading and maintenance doses will be based on participants' body weight per approved dose regimen.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The primary purpose of this study is to assess the safety, efficacy, pharmacokinetics, and pharmacodynamics of ravulizumab in participants who are prescribed and are receiving a higher than approved dose of eculizumab to treat paroxysmal nocturnal hemoglobinuria (PNH).

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented diagnosis of PNH, confirmed by high-sensitivity flow cytometry evaluation of red blood cells and white blood cells, with granulocyte or monocyte clone size of ≥ 5%.
2. Received 1200 mg eculizumab every 12 to 16 days (every 2 weeks) for at least 3 months prior to Screening.
3. LDH ≤ 2 x upper limit of normal (ULN) according to central laboratory, at Screening.
4. To reduce the risk of meningococcal infection (Neisseria meningitidis), all participants must be vaccinated against meningococcal infections within 3 years prior to initiating study drug.
5. Body weight ≥ 40 kilograms.

Key Exclusion Criteria:

1. History of major adverse vascular events within 6 months of Day 1.
2. History of bone marrow transplantation.
3. Lymphoma, leukemia, myelodysplastic syndrome, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
4. Concomitant use of anticoagulants is prohibited if not on a stable regimen for at least 2 weeks prior to Day 1.
5. Concomitant use of any of the following medications and not on a stable regimen (as judged by the Investigator) for the time period indicated prior to Screening:

   * Erythropoietin or immunosuppressants for at least 8 weeks
   * Systemic corticosteroids for at least 4 weeks
   * Vitamin K antagonists (for example, warfarin) with a stable international normalized ratio level for at least 4 weeks
   * Iron supplements or folic acid for 4 weeks
6. Live vaccine(s) within 1 month prior to Screening or plans to receive such vaccines during the study.
7. More than 1 LDH value > 2 × ULN within the 6 months prior to Day 1.
8. Platelet count < 30,000/cubic millimeter (30 × 10^9/Liter [L]) at Screening.
9. Absolute neutrophil count < 500/microliter (0.5 × 10^9/L) at Screening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Clinical Study Site, Leeds
  - Research Site, Leeds
  - Clinical Study Site, London
  - Research Site, London

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-PNH-401&attachmentIdentifier=f4f63037-1e40-4456-96df-06b466412244&fileName=ALXN1210-PNH-401-_CSR_synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a Screening Period of approximately 3 months and a Treatment Period of 351 days. Eligible participants were administered eculizumab 1200 milligrams (mg) every 2 weeks (q2w) optionally at home at the discretion of the Investigator, and preference of the participant during the Screening Period.
Groups:
- Ravulizumab: Participants received a loading dose of ravulizumab on Day 1 and maintenance treatment with ravulizumab on Day 15 and every 8 weeks (q8w) thereafter until Day 351. Ravulizumab loading and maintenance doses were based on the participant's body weight measured at the prior visit, per approved dosing regimen.
Period: Overall Study
Arm/Group | Ravulizumab
Started | 18
Received at Least 1 Dose of Study Drug | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received at least 1 dose of ravulizumab.
Groups:
- Ravulizumab: Participants received a loading dose of ravulizumab on Day 1 and maintenance treatment with ravulizumab on Day 15 and q8w thereafter until Day 351. Ravulizumab loading and maintenance doses were based on the participant's body weight measured at the prior visit, per approved dosing regimen.
Arm/Group | Ravulizumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.34) [lower limit 11.34]
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 0
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 15
  From 65-84 years | 3
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Free C5-associated BTH
Description: Free C5-associated BTH was defined as BTH concurrent with free C5 concentrations ≥0.5 micrograms (μg)/milliliter (mL). BTH was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin <10 grams {g}/deciliter {dL}], major adverse vascular event [MAVE], including thrombosis, dysphagia, or erectile dysfunction) in the presence of elevated lactate dehydrogenase (LDH) ≥2 * upper limit of normal (ULN).
Time Frame: Baseline through Day 351
Population: The FAS included all participants who received at least 1 dose of ravulizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 18
percentage of participants | 0 (0) [0 to 18.5]

2. Secondary Outcome: Percentage of Participants Who Experienced BTH
Description: BTH was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin <10 g/dL], MAVE, including thrombosis, dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2 * ULN.
Time Frame: Baseline through Day 351
Population: The FAS included all participants who received at least 1 dose of ravulizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 18
percentage of participants | 5.6 (0.1) [0.1 to 27.3]

3. Secondary Outcome: Percent Change From Baseline in LDH at Day 351
Time Frame: Baseline, Day 351
Population: The FAS included all participants who received at least 1 dose of ravulizumab. Here, 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ravulizumab
Number analyzed (Participants) | 14
percent change | -0.81 (6.132) [lower limit 6.132]

4. Secondary Outcome: Percentage of Participants Who Received a Red Blood Cell (RBC) Transfusion
Time Frame: Baseline through Day 351
Population: The FAS included all participants who received at least 1 dose of ravulizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 18
percentage of participants | 33.3 (13.3) [13.3 to 59.0]

5. Secondary Outcome: Percentage of Participants With Stabilized Hemoglobin
Description: Stabilized hemoglobin was defined as avoidance of a ≥2 g/dL decrease in hemoglobin level from baseline in the absence of transfusion from Baseline to Day 351.
Time Frame: Baseline through Day 351
Population: The FAS included all participants who received at least 1 dose of ravulizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 18
percentage of participants | 61.1 (35.7) [35.7 to 82.7]

ADVERSE EVENTS:
Time Frame: Baseline through Day 351
Description: Safety set included all participants who received at least 1 dose of ravulizumab.
Arm/Group | Ravulizumab
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ravulizumab (N=18)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ravulizumab (N=18)
Fatigue (General disorders) | 6 (8)
Non-cardiac chest pain (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (3)
Herpes zoster (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 3 (3)
Body temperature abnormal (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Extravascular haemolysis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT04320602/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT04320602/SAP_001.pdf